CLINICAL TRIAL: NCT03872791
Title: A Phase Ib/II Study to Evaluate Efficacy, Safety and Tolerability of KN046 Monotherapy or in Combination With Nab-paclitaxel in Subjects With Triple-negative Breast Cancer
Brief Title: A Study of KN046 in Subjects With Locally Advanced or Metastatic Triple-negative Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jiangsu Alphamab Biopharmaceuticals Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: KN046-203
Record Dates: First submitted 2019-03-07; First posted 2019-03-13 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-06

CONDITIONS: Triple-negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KN046 (Experimental): Subjects will receive KN046 at a dose of 3 mg/kg or 5 mg/kg via intravenous infusion on Days 1 and 15 of every 28-day cycle until disease progression, unacceptable toxicity or completion of 2 years of treatment
  Interventions: Biological: KN046
- KN046 plus nab-paclitaxel (Experimental): Subjects will receive KN046 at a dose of 3 mg/kg or 5 mg/kg via intravenous infusion on Days 1 and 15 of every 28-day cycle until disease progression, unacceptable toxicity or completion of 2 years of treatment Subjects will receive nab-paclitaxel at a dose of 100 mg/m2 via intravenous infusion on Days 1, 8 and 15 of every 28-day cycle until disease progression or unacceptable toxicity
  Interventions: Biological: KN046; Drug: Nab-paclitaxel

INTERVENTIONS:
Biological: KN046 — KN046 at a dose level of 3 or 5 mg/kg via intravenous infusion on Days 1 and 15 of 28-day cycle
Drug: Nab-paclitaxel — Nab-paclitaxel at dose level of 100 mg/m2 via intravenous infusion on Days 1, 8 and 15 of 28-day cycle
  Arms: KN046 plus nab-paclitaxel

SUMMARY:
This is an open-label, phase Ib/II, multi-center study to evaluate efficacy and safety of KN046 alone or in combination with nab-paclitaxel in subjects with locally advanced unresectable or metastatic triple negative breast cancer (TNBC). The study is composed of dose escalation and expansion parts. Every subject will subject tumor tissue used for biomarker evaluation. Each subject will receive KN046 or in combination with nab-paclitaxel untill confirmed progressive disease, unacceptable toxicity or withdrawal of informed consent whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent;
* Age of 18 or above;
* Histology confirmed locally advanced unresectable or metastatic triple-negative breaset cancer;
* (KN046 monotherapy) failed at least one prior anthracycline and taxane containing systemic treatment, (KN046 plus nab-paclitaxel) systemic treatment naive;
* Measurable disease at baseline;
* ECOG 0-1;
* Adequate organ functions.

Exclusion Criteria:

* Untreated active CNS metastasis or leptomeningeal metastasis;
* Subjects receiving immunosuppressive agents (such as steroids) for any reason should be tapered off these drugs before initiation of trial treatment;
* Has interstitial lung disease, or a history of pneumonitis that required oral or intravenous glucocorticoids to assist with management;
* Active autoimmune disease that might deteriorate when receiving an immunostimulatory agent; History of uncontrolled intercurrent illness; Known severe hypersensitivity reactions to antibody drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2019-05-30 (Actual); Primary Completion 2022-08-16 (Actual); Study Completion 2022-10-27 (Actual)

PRIMARY OUTCOMES:
IRC assessed objective response | From Day 1 to PD, assessed up to 12 months after last patient last dose
  Objective response is defined as complete response (CR) or partial response (PR), as determined by the independent review committee using RECIST v1.1 criteria. CR is defined as the disappearance of all TLs and SA reduction to less than (<) 10mm for nodal TLs/ non-TLs. PR is defined as >/=30% decrease in SD of TLs, taking as reference the baseline SD
IRC assessed duration of response | From Day 1 to PD, assessed up to 12 months after last patient last dose
  Duration of response is defined as the time period from the date of initial independent review committee assessed CR or PR until the date of PD or death from any cause, whichever occurs first. CR is defined as the disappearance of all TLs and SA reduction to <10mm for nodal TLs/ non-TLs. PR is defined as >/=30% decrease in SD of TLs, taking as reference the baseline SD. PD is defined as >/=20% relative increase and >/=5 mm of absolute increase in the SD of TLs, taking as reference the smallest SD recorded since treatment started, or appearance of 1 or more new lesions

SECONDARY OUTCOMES:
PFS rate at 6 and 12 months | From Day 1 to disease progression (PD) or death from any cause, assessed up to 12 months after last patient last dose
  PFS is defined as the time from Day 1 to the first occurrence of PD, as determined by the independent review committee or investigator using RECIST v1.1, or death from any cause during the study, whichever occurs first. PD is defined as greater than or equal to (>/=) 20 percent (%) relative increase and >/=5 millimeter (mm) of absolute increase in the sum of diameters (SD) of target lesions (TLs), taking as reference the smallest SD recorded since treatment started, or appearance of 1 or more new lesions. PFS rate at 6 and 12 months is defined as percentage of subjects who are alive without progressive disease or death at 6 and 12 months
Frequency and severity of treatment emergent adverse events | From Day 1 to 90 days after last dose of KN046, through study completion, an average of 1 year
  Treatment emergent adverse event is defined as those events with onset days occurring during the on-treatment period till 90 days after last dose of KN046 or if the worsening of an event is during the on-treatment period till 90 days after last dose of KN046
Percentage of subjects with anti-drug antibodies | Day 1 (pre-dose) to 90 days after last dose of KN046, through study completion, an average of 1 year
  ADA is defined as human anti-drug antibodies

CONTACTS AND LOCATIONS:
Locations (12):
- China (12):
  - National Cancer Center/Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Hunan Cancer Hospital, Changsha, Hunan
  - Nantong Tumor Hospital, Nantong, Jiangsu
  - JiLin Cancer Hospital, Changchun, Jilin
  - Liaoning Cancer Hospital, Shenyang, Liaoning
  - LiaoCheng People's Hospital, Liaocheng, Shandong
  - Zibo Municipal Hospital, Zibo, Shandong

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 6 months after publication
Access Criteria: Health care professionals or researches may raise request to Sponsor to have access to study report, sub-group analysis